CLINICAL TRIAL: NCT02654691
Title: DOLORISK: Understanding Risk Factors and Determinants for Neuropathic Pain - Chronic Neuropathy Following Chemotherapy
Brief Title: Chronic Neuropathy Following Chemotherapy
Acronym: DOLORISKCIPN
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Collaborators: University of Oxford (Other); Imperial College London (Other); University of Dundee (Other); Mentis Cura (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Kiel (Other); Lund University (Other); Technion, Israel Institute of Technology (Other); University Ghent (Other); Neuroscience Technologies S.L.P (Industry)
Responsible Party: Sponsor
Other Study IDs: CIPN-2015
Record Dates: First submitted 2015-12-22; First posted 2016-01-13 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Nervous System Diseases; Chronic Pain
Keywords: Chemotherapy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a clinical study which is a follow-up of a previous prospective questionnaire study. All patients who previously participated in the study will receive a new questionnaire and will be invited for a clinical examination.

DETAILED DESCRIPTION:
This is a clinical study which is a follow-up of a previous prospective questionnaire study. All patients who previously participated in the study will receive a new questionnaire and will be invited for a clinical examination. This is a collaboration and part of the data will be combined with other data in this collaboration

ELIGIBILITY:
Inclusion Criteria:

* all patients who have participated in a prospective questionnaire study

Exclusion Criteria:

* Not able to visit in person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent chemotherapy for a high-risk mamma-cancer and a high-risk colon-cancer from the period of 2011-2012 and who participated in a prospective questionnaire study (Ventzel et al. 2015).
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine J Bennedsgaard, MD, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Data is shared among collaborators (DOLORisk consortium)

REFERENCES:
- [Background] Ventzel L, Jensen AB, Jensen AR, Jensen TS, Finnerup NB. Chemotherapy-induced pain and neuropathy: a prospective study in patients treated with adjuvant oxaliplatin or docetaxel. Pain. 2016 Mar;157(3):560-568. doi: 10.1097/j.pain.0000000000000404. PMID 26529271
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Patients treated with docetaxel or oxaliplatin.
Period: Overall Study
Arm/Group | Chemotherapy
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 63

OUTCOME MEASURES:

1. Primary Outcome: Chemotherapy-induced Peripheral Neuropathy
Description: For case definition of neuropathy, The Toronto classification (Tesfaye et al. 2010) will be used.
  Numbers indicate confirmed neuropathy.
Time Frame: 5-year follow-up
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
participants | 21

2. Primary Outcome: Chemotherapy-induced Neuropathic Pain
Description: Neuropathic pain grading system. Neuropathic pain was graded as "possible", "probable", or "definite" in accordance with the NeuPSIG grading system (Pascal M et al, Wellcome Open Research 2018).
Time Frame: 5-year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
Participants | 19

3. Secondary Outcome: Sensory Abnormalities After Chemotherapy Assessed With Quantitative Sensory Testing (QST).
Description: Modified German Research Network on Neuropathic Pain QST protocol assessed sensory abnormalities after chemotherapy assessed with quantitative sensory testing (QST).
Time Frame: 5-year follow-up
Population: Patients with an abnormal value indicating loss of function
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 62
participants
  Abnormal thermal detection | 11
  Abnormal vibration detection | 18
  Abnormal mechanical detection threshold | 11
  Abnormal paradoxical heat sensation | 16
  Abnormal mechanical pain threshold | 8

4. Secondary Outcome: Neuronal Excitability Changes After Chemotherapy Assessed With Threshold Tracking: Sensory
Description: Measurements found with threshold tracking. The most common sensory parameters assessed with sensory threshold tracking. Outcomes are extracted from the QTrack software. The relative refractory period (RRP) is the interval of time during which a second action potential can be initiated, refractoriness is change in threshold by a preceding simple impulse, and specifically at 2,5 ms. A shorten RRP makes the nerve more excitable and longer RRP less excitable (values see result 21 for refractoriness at 2.5 ms, superexcitability and subexcitability).
Time Frame: 5-year follow-up
Population: Sensory recordings from participants, the relative refractory period
Measure: Mean (Standard Error); unit: ms
Arm/Group | Chemotherapy
Number analyzed (Participants) | 55
ms | 3.1 (1.0)

5. Secondary Outcome: Anxiety and Depression Using the Patient Reported Outcomes Measurement Information System (PROMIS).
Description: Number of patients with mild, moderate or severe symptoms of depression or anxiety. Patient Reported Outcomes Measurement Information System (PROMIS) used to assess if the patients has a mild, moderat or severe symptoms of depression/anxiety. The scores from the questionnaires were converted into T-scores, which were used in grading the patients with mild , moderate or severe symptoms of depression or anxiety. A higher score indicates worse outcome. The minimum is no depression or anxiety and the maximum is severe depression or anxiey. Mild: T-score ≥55 and <65 Moderate: ≥65 and <75 Severe ≥75
Time Frame: 5-year follow-up
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
participants
  Anxiety | 12
  Depression | 12
  Anxiety or Depression | 16

6. Secondary Outcome: Anxiety and Depression Using the Hospital Anxiety and Depression Scale (HADS).
Description: Mean scores using HADS of all participants. The score for anxiety and depression indicate the sum of 7 questions, each graded from 0 to 3. This means that a person can score between 0 (minimum) and 21 (maximum) for either anxiety or depression. Higher score meaning more symptoms of a possible depression or anxiety.
Time Frame: 5-year follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
score on a scale
  Anxiety | 4.38 (3.76)
  Depression | 2.40 (2.34)

7. Secondary Outcome: Fatigue Using the Patient Reported Outcomes Measurement Information System (PROMIS).
Description: Number of patients with mild, moderate or severe fatigue. PROMIS used to assess if the patients has a mild, moderat or severe symptoms of fatique. The scores from the questionnaires were converted into T-scores, which were used in grading the patients with mild, moderate or severe symptoms of fatigue. The minimum is no fatigue (T-score<50) and maximum severe fatigue (T-score ≥75). Higher scores mean a worse outcome. Mild: T-score ≥55 and <65 Moderate: ≥65 and <75 Severe ≥75
Time Frame: 5-year follow-up
Population: Numbers given is patients with mild, moderate or severe fatigue.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
Participants | 25

8. Secondary Outcome: Quality of Life Using EuroQol (EQ-5D).
Description: The participants were asked to provided a score from 1-100 regarding quality of life on the Quality of life using EuroQol (EQ-5D). Minimum score 0, maximum score 100. A higher score indicate better outcome
Time Frame: 5-year follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
units on a scale | 78.4 (17.2)

9. Secondary Outcome: Personality Using the 10-item Personality Inventory (TIPI).
Description: The Personality using the 10-item Personality Inventory (TIPI). TIPI is divided in 5 parameters Extraversion, Agreeableness, Conscientiousness, Emotional Stability, Openness. Minimum value is 2 and maximum value i 14. Higher scores indicate more Openness, Conscientiousness, Extraversion, Agreeableness and Emotional Stability
Time Frame: 5-year follow-up
Population: Answers are missing for 1 participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 62
units on a scale
  Extraversion | 4.5 (1.5)
  Agreeableness | 4.9 (1.1)
  Conscientiousness | 5.2 (1.1)
  Emotional Stability | 5.2 (1.3)
  Openness | 5.3 (1.1)

10. Secondary Outcome: Personality Using the International Personality Item Pool (IPIP).
Description: Personality using the International Personality Item Pool (IPIP). A score were given from answering 10 questions regarding emotionel stability. Each question has 5 possible answers from 1 very inaccuate to 5 very accurate. Minimum combined value 10, maximum combined value 50. Higher score indicates worse outcome.
Time Frame: 5-year follow-up
Population: Results from 1 participant were missing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 62
score on a scale | 34.3 (7.6)

11. Secondary Outcome: Pain Catastrophizing Using the Pain Catastrophizing Scale(PCS).
Description: Participants answered 13 question, which were each graded on a scale from 0-4 and combined to a sum scale.. The results are a mean score for all participants. The minimum value is 0 and the maximum value is 72. Higher scores indicate more Pain catastrophizing.
Time Frame: 5-year follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
score on a scale | 7.6 (9.4)

12. Secondary Outcome: Morphology of Small Fibers in Cornea After Chemotherapy by Corneal Confocal Microscopy (CCM).
Description: The fibers in the cornea were scanned in one eye with the Heidelberg Retina Tomograph III laser-scanning confocal microscope (Heidelberg Engineering GmbH, Heidelberg, Germany). An automatic programme calculated the cornea nerve branches density (CNBD) and the cornea nerve fiber density (CNFD).
Time Frame: 5-year follow-up
Population: Missing data in 10 patients
Measure: Mean (Standard Deviation); unit: units/mm2
Arm/Group | Chemotherapy
Number analyzed (Participants) | 53
units/mm2
  CNBD | 30.5 (13.5)
  CNFD | 22.8 (7.8)

13. Secondary Outcome: Blood Samples DNA
Description: Numbers indicate the number of participants, who had a blood sample collected. Potential gene associations in the development of painful neuropathy will be assessed together with other samples in the DOLORisk collaboration. The results here present the number of subjects who had a DNA blood sample taken.
Time Frame: 5-year follow-up
Population: Numbers indicate the number of participants, who had a blood sample collected. Not analyzed separately
Measure: Number; unit: participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
participants | 58

14. Secondary Outcome: Pain Interference by Patient Reported Outcomes Measurement Information System (PROMIS).
Description: Numbers given is patients with mild, moderate or severe pain interference of the patients with neuropathic pain. Patient Reported Outcomes Measurement Information System PROMIS used to assess if the patients has a mild, moderate or severe symptoms of pain interference. The scores from the questionnaires were converted into T-scores, which were used in grading the patients with mild, moderate or severe pain interference. The mimimum is no interference (T-score <50) and maximum is Severe (T-score≥70)). Severe indicated more interference
Time Frame: 5-year follow-up
Population: Of the 63 included in the study, 19 patients had symptoms of neuropathic pain. Numbers given is patients with mild, moderate or severe pain interference of the patients with neuropathic pain.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 19
Participants | 17

15. Secondary Outcome: Pain Descriptors by Douleur Neuropathique 4 (DN4).
Description: number of participants with a possible painful neuropathy with the Douleur Neuropathique 4DN4. Yes/no questions regarding symptoms and signs of neuropathic pain. In total the participants answered 7 questions. Each question is a yes or no and are combined to a sum score of number of positive answers. Minimum score is 0 and maximum score is 7. Higher score indicates larger probability of neuropathic Pain. A score of 3 or above indicates a possible painful neuropathy.
Time Frame: 5-Year follow-up
Population: Of the 63 included in the study, 19 patients had symptoms of neuropathic pain. The result are the number of participants with a possible painful neuropathy with the DN4.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 19
Participants | 13

16. Secondary Outcome: Pain Descriptors by Neuropathic Pain Symptom Inventory (NPSI).
Description: The results were given on a scale from 0-100 for each of the 5 dimensions on the Neuropathic Pain Symptom Inventory (NPSI). Higher scores indicate worse symptoms. The sum score is the sum divided by 5. Minimum score is 0 and maximum score is 100.
Time Frame: 5-Year follow-up
Population: Of the 63 included in the study, 19 patients had symptoms of neuropathic pain. The result are the score of participants with a neuropathic pain.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 19
score on a scale | 23.3 (20.9)

17. Secondary Outcome: Neuropathy Using the Toronto Clinical Scoring System (TCSS).
Description: The Toronto Clinical Scoring System(TCSS), grades the severity of neuropathy and consists of 6 questions with the presence and description of symptoms and a 7-item clinical examination with reflexes in the lower extremities and a bedside sensory testing with pinprick, vibration, temperature, light touch and position of the 1st toe. The score ranges from 0-19. Higher score indicate worse outcome.
Time Frame: 5-year follow-up
Population: Results wer missing in 4 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 59
score on a scale | 4.8 (3.2)

18. Secondary Outcome: Neuropathy Using the Total Neuropathy Score.
Description: The TNScompact consists of 7 questions regarding sensory symptoms, motor symptoms, autonomic symptoms, pin sensation, vibrations sensitivity, strength and tendon reflexes graded from 0-4. The scores are combined and thus 0 being the lowest score possible and 28 being the highest score possible. A high score indicate severe neuropathy.
Time Frame: 5-year follow-up
Population: The results were missing for 5 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy
Number analyzed (Participants) | 58
score on a scale | 3.9 (3.0)

19. Secondary Outcome: Neuropathy Using the Michigan Neuropathy Screening Instrument (MNSI).
Description: A cut-off ≥ 4/13 abnormal responses has been suggested as the cut-off to define polyneuropathy.
Time Frame: 5-year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 63
Participants | 21

20. Secondary Outcome: Neuronal Excitability Changes After Chemotherapy Assessed With Threshold Tracking: Motor
Description: Measurements found with threshold tracking. The most common motor parameters assessed with threshold tracking. Outcomes are extracted from the QTrack software. The relative refractory period (RRP) is the interval of time during which a second action potential can be initiated, refractoriness is change in threshold by a preceding simple impulse, and specifically at 2,5 ms. A shorten RRP makes the nerve more excitable and longer RRP less excitable (values see result 22 for refractoriness at 2.5 ms, superexcitability and subexcitability).
Time Frame: 5-year follow-up
Population: Motor recordings from participants, relative refractory period
Measure: Mean (Standard Error); unit: ms
Arm/Group | Chemotherapy
Number analyzed (Participants) | 60
ms | 3.0 (1.0)

21. Secondary Outcome: Neuronal Excitability Changes After Chemotherapy Assessed With Threshold Tracking: Sensory
Description: Measurements found with threshold tracking. The most common sensory parameters assessed with sensory threshold tracking. Outcomes are extracted from the QTrack software. The relative refractory period (RRP) is the interval of time during which a second action potential can be initiated, refractoriness is change in threshold by a preceding simple impulse, and specifically at 2,5 ms. A shorten RRP makes the nerve more excitable and longer RRP less excitable (values see result 21 for refractoriness at 2.5 ms, superexcitability and subexcitability). Superexcitability and subexcitablity are measured in the recovery period. The recovery cycle is characterized by changes in axonal excitability following a supramaximal conditioning stimulus. The cycle includes a relative refractory period (at short inter-stimulus intervals), superexcitable period (when the threshold is reduced), and subexcitable period (when the nerve is less excitable).
Time Frame: 5-year follow-up
Population: Sensory recordings from participants, refractoriness at 2.5 ms, superexcitability and subexcitability
Measure: Mean (Standard Error); unit: percentage of 100%
Arm/Group | Chemotherapy
Number analyzed (Participants) | 55
percentage of 100%
  Refractoriness at 2.5 ms | 11.0 (1.9)
  Superexcitability | 17.4 (0.8)
  Subexcitability | 10.9 (0.8)

22. Secondary Outcome: Neuronal Excitability Changes After Chemotherapy Assessed With Threshold Tracking: Motor
Description: Measurements found with threshold tracking. The most common motor parameters assessed with threshold tracking. Outcomes are extracted from the QTrack software. The relative refractory period (RRP) is the interval of time during which a second action potential can be initiated, refractoriness is change in threshold by a preceding simple impulse, and specifically at 2,5 ms. A shorten (RRP) makes the nerve more excitable and longer RRP less excitable (values see result 22 for refractoriness at 2.5 ms, superexcitability and subexcitability). Superexcitability and subexcitablity are measured in the recovery period. The recovery cycle is characterized by changes in axonal excitability following a supramaximal conditioning stimulus. The cycle includes a relative refractory period (at short inter-stimulus intervals), superexcitable period (when the threshold is reduced), and subexcitable period (when the nerve is less excitable).
Time Frame: 5-year follow-up
Population: Motor recordings from participants, refractoriness at 2.5 ms, superexcitability and subexcitability
Measure: Mean (Standard Error); unit: percentage of 100%
Arm/Group | Chemotherapy
Number analyzed (Participants) | 60
percentage of 100%
  Refractoriness at 2.5 ms | 18.8 (1.9)
  Superexcitability | 21.8 (0.8)
  Subexcitability | 16.2 (0.7)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse events only measured during survey. There is no arm or group and no intervention.
Groups:
- Chemotherapy: There were no adverse events
Arm/Group | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT02654691/Prot_SAP_000.pdf